CLINICAL TRIAL: NCT03131128
Title: A Pilot Study of the Effectiveness of Mindfulness-based Intervention as a Workplace Health Promotion Program on Weight Loss
Brief Title: The Effectiveness of Mindfulness-based Intervention as a Workplace Health Promotion Program on Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Yeh, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ChungShanMU
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Mindfulness; Weight Loss; Workplace; Health Promotion
Keywords: Mindfulness-based intervention; Weight loss; Workplace health promotion; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: The workers with overweight or obesity provided by the company will be randomly assigned to Group A (by MBI) or Group B (by the intervention of health education).
Masking Description: The researchers will explain the purpose and steps of the study to all the participants and get their informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Intervention (Experimental): 2 sessions of diet nutrition education and 6 sessions of Mindfulness-based intervention, 1.5 hours each session.
  Interventions: Behavioral: Mindfulness-based Intervention
- Health Education Intervention (Active Comparator): 2 sessions of diet nutrition education and 6 sessions of Health Education, 1.5 hours each session.
  Interventions: Behavioral: Health Education Intervention

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention — 1. Keeping mindful when selecting food.
  2. Be aware of hunger and satiety by the body clues.
  3. Understanding how stress affect diet and life, and learn how to cope with stress in life.
  4. Learning to identify overeating caused by mood, social stress and specific food.
  Arms: Mindfulness-based Intervention
Behavioral: Health Education Intervention — 1. Identifying improper diet patterns and attitudes
  2. Understanding the impact of irrational cognition and attitudes on dietary behavior
  3. Training coping skills for stresses in real life and preventing the recurrence of bulimia.
  Arms: Health Education Intervention

SUMMARY:
The present study will carry out a workplace health promotion via MBI with lessons of dietary behavior to help overweight or obese workers to loss weight.

DETAILED DESCRIPTION:
The study will adopt a longitudinal research design with randomized quasi- experimental trial. The workers with overweight or obesity (BMI≧24) provided by the company will be randomly assigned to Group A (four lessons of dietary behavior and six lessons of MBI) or Group B (four lessons of dietary behavior and six lessons of mental health). There will be 100 participants in each group. Data will be collected five times. The research questionnaire includes basic information (including BMI, waist circumference, etc), Perceived Stress Scale, The Five Facet Mindfulness Questionnaire, Food Cravings Questionnaire, the scale of physical activity and information regarding dietary behavior.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 20 to 65 years old;
2. full-time workers with BMI ≧ 24;
3. motivated to participate in the study;

Exclusion Criteria:

1. suffering from mental illness or in an acute episode;
2. suffering from life threatening or other major physical illness;
3. no motivation to participate in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Up to 10 months
  Body weight will be recorded during the study carried out.

SECONDARY OUTCOMES:
Dietary Behavior | Up to 10 months
  Using the Dietary Behavior Questionnaire to measure the intake of types and proportion of food.
Food Cravings | Up to 10 months
  Measuring the level of food cravings, use the Likert six-point scoring method, from 1-6 points, a total of 21 questions. The higher scores indicate higher food cravings levels.
Perceived Stress | Up to 10 months
  Measuring the level of perceived stress, using the Likert five-point scoring method, from 0-4 points, a total of 10 questions .The higher scores indicate higher pressure levels.
The level of Mindfulness | Up to 10 months
  Measuring the level of Mindfulness, using the Likert five-point scoring method, a total of 39 questions, including the five concepts, namely: awareness (8 questions), description (8 questions), non-judging (8 questions), observation (8 questions), and non-reaction (7 questions). The higher scores indicate higher levels of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Cheng Tang, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No